CLINICAL TRIAL: NCT06188468
Title: ImmunoPET Targeting Trophoblast Cell-surface Antigen 2 (Trop-2) in Solid Tumors and Compared with 18F-FDG
Brief Title: ImmunoPET Targeting Trophoblast Cell-surface Antigen 2 (Trop-2) in Solid Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: XMYY-2024KY024
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Tumor; Solid Tumor; Positron-Emission Tomography
Keywords: Tumor; Solid; Positron-Emission Tomography; Trop-2; Diagnosis
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 68Ga-MY6349 (Experimental): Each subject receives a single intravenous injection of 68Ga-MY6349 and undergoes PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: standard-of-care imaging (18F-FDG, 68Ga-PSMA, or 68Ga-DOTATATE PET/CT), 68Ga-MY6349 PET/CT

INTERVENTIONS:
Diagnostic Test: standard-of-care imaging (18F-FDG, 68Ga-PSMA, or 68Ga-DOTATATE PET/CT), 68Ga-MY6349 PET/CT — Each subject receives a single intravenous injection of standard-of-care imaging radiopharmaceuticals (18F-FDG, 68Ga-PSMA, or 68Ga-DOTATATE) and 68Ga-MY6349, and undergoes PET/CT imaging within the specified time.

SUMMARY:
The objective of the study is to construct a noninvasive approach 68Ga-MY6349 PET/CT to detect the Trop-2 expression of tumor lesions in patients with solid tumors and to identify patients benefiting from Trop-2 targeting antibody-drug conjugate treatment.

DETAILED DESCRIPTION:
As a new trophoblast cell-surface antigen 2 (Trop-2) targeting PET radiotracer, 68Ga-MY6349 is promising as an excellent imaging agent applicable to various cancers. In this research, subjects with various types of tumors underwent contemporaneous 68Ga-MY6349 and standard-of-care imaging (18F-FDG, 68Ga-PSMA, or 68Ga-DOTATATE PET/CT) either for an initial assessment or for recurrence detection. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The numbers of positive tumor lesions of standard-of-care imaging and 68Ga-MY6349 PET/CT were recorded by visual interpretation. The diagnostic accuracy of 68Ga-MY6349 was calculated and compared to standard-of-care imaging.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (aged 18 years or older);
2. patients with suspected or newly diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report);
3. patients who had scheduled both standard-of-care imaging (18F-FDG, 68Ga-PSMA, or 68Ga-DOTATATE PET/CT) and 68Ga-MY6349 PET/CT scans;
4. patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

1. patients with pregnancy;
2. the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluate the feasibility of PET/CT imaging with 68Ga-MY6349 for the non-invasive assessment of Trop2 expression in various cancer types. | 1 week
  Tumor Trop2 expression analysis in a fresh biopsy sample will be correlated to 68Ga-MY6349 tumor uptake, evaluated by measuring standardized uptake value (SUV) on the 68Ga-MY6349 PET/CT.

SECONDARY OUTCOMES:
To investigate the superiority of 68Ga-MY6349 PET/CT over 18F-FDG PET/CT in some tumors through comparative analysis | 2 weeks
  The numbers of positive primary and metastatic lesions of standard-of-care imaging (18F-FDG PET/CT) and 68Ga-MY6349 PET/CT were recorded by visual interpretation.
Description of 68Ga-MY6349 uptake by measuring standardized uptake value (SUV) in various types of tumors | 1 week
  Standardized uptake value (SUV) of 68Ga-MY6349 PET/CT for each target lesion of subject or suspected primary tumor or/and metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

REFERENCES:
- [Derived] Chen H, Zhao L, Pang Y, Shi J, Gao H, Sun Y, Chen J, Fu H, Cai J, Yu L, Zeng R, Sun L, Wu H, Wang Z, Wang F. 68Ga-MY6349 PET/CT imaging to assess Trop2 expression in multiple types of cancer. J Clin Invest. 2024 Nov 7;135(1):e185408. doi: 10.1172/JCI185408. PMID 39509246